CLINICAL TRIAL: NCT02039102
Title: Use of Hormonal Contraceptives in Relation to Asthma and Wheezing Disorders in Scottish Women: a Population-based Cross-sectional Survey
Brief Title: Contraceptive Use and Respiratory Conditions Among Scottish Women
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 75764
Record Dates: First submitted 2014-01-15; First posted 2014-01-17 (Estimated); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Asthma
Keywords: hormonal contraceptives; combined pills; progesterone-only contraceptives; body mass index; asthma; Scotland; women
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non-users of hormonal contraceptives
- Users of hormonal contraceptives

SUMMARY:
Studies examining the sex differences in the epidemiology and morbidity patterns of asthma show that the rates of disease severity, healthcare utilisation, and poor quality of life are considerably higher in women than in men, and this has been attributed to endogenous and exogenous sex hormonal factors. Studies examining the impact of use of hormonal contraceptives on the risk of asthma and asthma-related conditions are few, yet findings are conflicting.

In the present study, the investigators utilize data from the Scottish Health Survey, a national representative sample, to investigate the associations between current use of hormonal contraceptives and the prevalence of self-reported doctor-diagnosed current asthma and wheezing symptoms in Scottish women. The investigators hypothesize that while current use of any hormonal contraceptives and combined oral pills are associated with higher prevalence of asthma and asthma outcomes, current use of progesterone-only contraceptives is not associated with asthma. A secondary aim of the current study is to examine whether there is evidence of any biological interaction between use of hormonal contraceptives and BMI in relation to the risk of asthma and asthma outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant
* Woman
* 16-45 years old

Exclusion Criteria:

* Pregnant
* Man
* Younger than 16 years or older than 45 years old

Ages: 16 Years to 45 Years | Sex: Female
Age Groups: Child, Adult
Study Population: Non-pregnant women aged 16-45 years
Sampling Method: Probability Sample
Enrollment: 3257 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Self-reported doctor-diagnosed current asthma | During the past 12 months

SECONDARY OUTCOMES:
Self-reported wheezing symptom | During the past 12 months
Self-reported current treatment for asthma/wheeze | During the past 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ediburgh, Edinburgh, United Kingdom

REFERENCES:
- [Background] Macsali F, Real FG, Omenaas ER, Bjorge L, Janson C, Franklin K, Svanes C. Oral contraception, body mass index, and asthma: a cross-sectional Nordic-Baltic population survey. J Allergy Clin Immunol. 2009 Feb;123(2):391-7. doi: 10.1016/j.jaci.2008.10.041. Epub 2009 Jan 3. PMID 19121863
- [Background] Lange P, Parner J, Prescott E, Ulrik CS, Vestbo J. Exogenous female sex steroid hormones and risk of asthma and asthma-like symptoms: a cross sectional study of the general population. Thorax. 2001 Aug;56(8):613-6. doi: 10.1136/thorax.56.8.613. PMID 11462063
- [Background] Salam MT, Wenten M, Gilliland FD. Endogenous and exogenous sex steroid hormones and asthma and wheeze in young women. J Allergy Clin Immunol. 2006 May;117(5):1001-7. doi: 10.1016/j.jaci.2006.02.004. PMID 16675325